CLINICAL TRIAL: NCT06025864
Title: Support Protocol for Face-to-face and Teleservice Breastfeeding for Puerperal Women and Mothers of Babies With Congenital Heart Disease: a Randomized Clinical Trial
Brief Title: Protocol to Support Breastfeeding for Postpartum Women and Mothers of Babies With Congenital Heart Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Collaborators: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Responsible Party: Principal Investigator, Fernanda Lucchese, Principal Investigator, Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5947.21
Record Dates: First submitted 2023-08-21; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Breastfeeding; Congenital Heart Disease
Keywords: breast milk; congenital heart desease; nutritional status; 6 months; call center
MeSH Terms: conditions — Breast Feeding; Heart Defects, Congenital | interventions — Lactation

STUDY DESIGN:
Intervention Model Description: Multicenter Randomized Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Support for breastfeeding and depletion of breast milk throughout the 6 months. Free and professional support through monthly consultations and videos on the subject.
  Interventions: Other: Breastfeeding
- Control Group (No Intervention): All mothers were followed up for 6 months and received a breastfeeding support booklet virtually, through a cell phone application. The booklet provides basic information about breastfeeding and possible complications. The recruited mothers also received a notebook to record the date, duration, volume and frequency of breastfeeding and/or milk collections, and the use of alternative routes such as a bottle, cup or enteral nutrition. At the initial visit, all mothers were given a standard measuring cup to measure the volume of milk used up in the household each day.
  In addition, all mothers received a call 7 days after delivery to apply the Portuguese version of the Breastfeeding Self-Efficacy Survey - Short Form: BSES-SF. This questionnaire was reapplied after 90 days.

INTERVENTIONS:
Other: Breastfeeding — Over the 6 months of the intervention, 1 video per month was sent, a total of 6 videos, via the mobile application, with guidance on breastfeeding: the importance of maternal hydration; myths and truths about the mother's diet; practical guidance on breastfeeding; baby's gastric capacity; picking up and positioning the baby during breastfeeding and storing milk for the return to work. There were also 1 call per month, with an average duration of 15 minutes, with a breastfeeding consultant nutritionist, aiming to solve doubts and difficulties that month. In order to provide complete assistance, virtual groups were created via the WhatsApp application, with a nutritionist and a health academic to solve doubts, provide emotional support and exchange information when necessary.
  According to the region or municipality of origin of the mother-baby dyad, when necessary, this study provided the loan of a breast pump during the follow-up period or 6 months.
  Arms: Intervention Group

SUMMARY:
To evaluate the effect of applying a hybrid protocol (face-to-face and via call center) of breastfeeding assistance and guidance on the duration of breast milk supply to babies with congenital heart disease for 6 months.

DETAILED DESCRIPTION:
The objective of this randomized, multicenter clinical trial is to evaluate the effect of applying a hybrid protocol (face-to-face and telemarketing) of assistance and guidance on breastfeeding and duration of breast milk supply for infants with congenital heart disease in the first 6 months of life. Recruitment of infants diagnosed with congenital heart disease occurs within the first 72 hours of life, being followed up for 6 months.

Initially, the mothers in the control group, as well as the mothers in the intervention group, receive a booklet with guidelines on breastfeeding, a standardized measuring cup for milk collections and a breastfeeding booklet.

In addition, mothers in the intervention group receive monthly videos with guidance on breastfeeding, monthly consultations with a breastfeeding consultant and a support group via whatsapp with the researcher and scientific initiation student until the baby is 6 months old.

ELIGIBILITY:
Inclusion Criteria:

* Infants diagnosed with congenital heart disease,
* The parents must have a cell phone enabled to receive video calls.

Exclusion Criteria:

* Mothers carriers of the human immunodeficiency virus (HIV),
* Mothers users of medications without medical indication to initiate or maintain breastfeeding.

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
Breast milk supply rate during the baby's 6-month period | Up to 6 months
  Increase milk supply directly from the mother's breast or through pumps for use in alternative routes.

SECONDARY OUTCOMES:
Compare the time of breastfeeding | Up to 6 months
  Compare the time of offering the breast between the control group and the intervention group
Breastfeeding self-efficacy before and during the intervention | Up to 6 months
  The breastfeeding self-efficacy questionnaire in a reduced format (BSES-SF) will be applied in two moments during the infant's 6 months of life, and the effectiveness of the interventions can be observed. The score can vary from 1 to 70, where higher results reflect greater self-efficacy in breastfeeding.
Assessment of the nutritional status of infants at 6 months of age using the growth curves of the World Health Organization and classified according to the Z score | Up to 6 months
  Assess the nutritional status of infants at 6 months of age through weight and height. These data will be placed on the nutritional assessment curves of the World Health Organization (WHO) and classified using the Z score. Afterwards, the results between the intervention and control groups will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Lucchese-Lobato, PHD, Principal Investigator — Instituto de Cardiologia de Porto Alegre
Locations (1):
- Juliana Caprini, Caxias do Sul, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carlsen EM, Kyhnaeb A, Renault KM, Cortes D, Michaelsen KF, Pryds O. Telephone-based support prolongs breastfeeding duration in obese women: a randomized trial. Am J Clin Nutr. 2013 Nov;98(5):1226-32. doi: 10.3945/ajcn.113.059600. Epub 2013 Sep 4. PMID 24004897
- [Result] Dodt RC, Joventino ES, Aquino PS, Almeida PC, Ximenes LB. An experimental study of an educational intervention to promote maternal self-efficacy in breastfeeding. Rev Lat Am Enfermagem. 2015 Jul-Aug;23(4):725-32. doi: 10.1590/0104-1169.0295.2609. PMID 26444176